CLINICAL TRIAL: NCT05176392
Title: Combined Nonpharmacological Therapies for MTBI-Related Headaches
Brief Title: Combined Transcranial Magnetic Stimulation and Therapy for MTBI Related Headaches
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CP200229; W81XWH2110831 (Other Grant/Funding Number: Department of Defense); H210076 (Other: VA San Diego Healthcare System)
Record Dates: First submitted 2021-11-24; First posted 2022-01-04 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: TBI (Traumatic Brain Injury); Headache; Depression
Keywords: rTMS; transcranial magnetic stimulation; therapy
MeSH Terms: conditions — Brain Injuries, Traumatic; Headache; Depression

STUDY DESIGN:
Intervention Model Description: Each participant will be randomized into one of 4 groups. Blocked randomization will be used with random block size of 4 or 8. Participants will be randomized to study groups in a 1:1:1:1 ratio.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participant, study coordinators and the investigators will be blinded to the rTMS treatment. The participant will be blinded to the therapy group (headache management or headache education).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active rTMS with telehealth headache management therapy (Active Comparator): Participants receive both active rTMS treatment at the left dorsolateral prefrontal cortex and therapy for headache management
  Interventions: Device: Active rTMS; Behavioral: Headache Management Therapy
- Active rTMS with telehealth headache education control (Other): Participants receive active rTMS treatment at the left dorsolateral prefrontal cortex and headache education
  Interventions: Device: Active rTMS; Behavioral: Headache Education Control
- Sham rTMS with telehealth headache management therapy (Other): Participants receive sham rTMS treatment at the left dorsolateral prefrontal cortex and therapy for headache management
  Interventions: Behavioral: Headache Management Therapy; Device: Sham rTMS
- Sham rTMS with telehealth headache education control (Sham Comparator): Participants receive sham rTMS treatment at the left dorsolateral prefrontal cortex and headache education
  Interventions: Device: Sham rTMS; Behavioral: Headache Education Control

INTERVENTIONS:
Device: Active rTMS — Active rTMS will be given at the left dorsolateral prefrontal cortex with a double blind TMS coil.
  Arms: Active rTMS with telehealth headache education control; Active rTMS with telehealth headache management therapy
Behavioral: Headache Management Therapy — Therapy will be provided on headache management.
  Arms: Active rTMS with telehealth headache management therapy; Sham rTMS with telehealth headache management therapy
Device: Sham rTMS — Sham rTMS will be given at the left dorsolateral prefrontal cortex. All parameters of the treatment will appear identical to the active treatment, with only the rTMS coil used to administer the treatment flipped 180 degrees to prevent stimulation.
  Arms: Sham rTMS with telehealth headache education control; Sham rTMS with telehealth headache management therapy
Behavioral: Headache Education Control — In the control, educational sessions on headaches will be provided.
  Arms: Active rTMS with telehealth headache education control; Sham rTMS with telehealth headache education control

SUMMARY:
This study will assess the combined effectiveness of repetitive transcranial magnetic stimulation (rTMS) and telehealth based therapy in helping manage mild traumatic brain injury (mTBI) related headaches. The investigators hypothesize that active rTMS combined with telehealth therapy will provide marked reduction in mTBI related headaches and symptoms in comparison to their placebo counterparts.

DETAILED DESCRIPTION:
This study will be enrolling a total of 240 veterans or active military over a 4 year period at the VA San Diego Healthcare System (VASDHS). Participants will be randomized into one of four groups:

Group A: active rTMS with telehealth headache management therapy Group B: active rTMS with telehealth headache education control Group C: sham rTMS with telehealth headache management therapy Group D: sham rTMS with telehealth headache education control

Individual participation will consist of 19 visits to the VASDHS and 11 telehealth sessions over the course of 6-7 months. The in person visits will be divided into the following phases:

1. PRE-TREATMENT ASSESSMENTS PHASE (weeks 1-2) which consists of Visit 1 (Screening Visit) and Visit 2 (Baseline Assessments with MRI scan);
2. INDUCTION TREATMENT PHASE (weeks 3-4) consists of Visits 3-12 (10 weekday neuronavigation guided rTMS sessions at >24 and <72 hours apart); and
3. POST-TREATMENT ASSESSMENTS AND MAINTENANCE TREATMENT PHASE (weeks 5-24) consists of 4 initial biweekly post-induction treatment assessments and maintenance treatments (Visits 13-16)) and two additional monthly post-induction assessments and maintenance treatments (Visits 17-18) and one final study visit (Visit 19).

Eight weekly telehealth therapy/education sessions will be conducted from week 3 to 10 with additional three bolster sessions at 4 weeks apart. During the baseline and follow up visits, assessments will be conducted to evaluate headaches, neurobehavioral symptoms, depressive symptoms, post-concussion symptoms, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Mild Traumatic Brain Injury (mTBI)
2. Chronic headaches > 3 months after injury
3. Aged 18-65
4. No prior TMS treatment
5. Persistent Headaches with an intensity > 30 / 100
6. No history of daily headache prior to mTBI

Exclusion Criteria:

1. Pregnant
2. Pacemaker or any metal in body that would prevent MRI
3. History of dementia or major psychiatric disease, such as bipolar disorder or schizophrenia
4. Presence of any other chronic neuropathic pain states
5. History of seizure
6. Pending litigation
7. Can't understand English
8. History of chronic headache like migraine prior to mTBI
9. Evidence in chart of exacerbation of depressive/anxiety symptoms, active substance dependence, suicidal intent or attempt within previous month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Intensity of Persistent Headaches | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Assesses the intensity of persistent headaches, from a scale of 0, being no pain, to 10, being worst possible pain.
Intensity of Debilitating Headaches | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Assesses the intensity of debilitating headaches, from a scale of 0, being no pain, to 10, being worst possible pain.
Persistent Headache Frequency | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Assesses the frequency per week of persistent headaches
Debilitating Headache Frequency | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Assesses the frequency per week of debilitating headaches
Debilitating Headache Interference | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Assesses the interference of debilitating headaches for activities of daily living, from 0, being no interference, to 10, being worst possible interference.

SECONDARY OUTCOMES:
Headache Impact Test | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Measures the impact of headache on an individual's ability to function at work, school, home, and/or social situations. Each item is measured from never, rarely, sometimes, very often, or always, with scores of 6, 8, 10, 11, and 13 respectively. A higher score correlates to a greater negative impact of headaches on quality of life.
Neurobehavioral Symptom Inventory | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Assesses the severity of symptoms in the following areas: somatic, cognitive, affective, and sensory. Each item ranges from 0-4 with a higher score indicating a worse outcome.
Hamilton Rating Scale for Depression | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Rates the severity of symptoms observed in depression such as low mood, insomnia, agitation, anxiety and weight loss. Scores range from 0 to 53, with a higher score indicating a larger degree of depression.
Rivermead Post-Concussion Symptoms Questionnaire | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Assesses somatic, cognitive, and emotional symptoms experiences after traumatic brain injury. Each item ranges from 0-4, with a higher score indicating a worse outcome.
Short Form Health Survey-36 | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Measures health status and quality of life in regards to eight main areas: vitality, physical functioning, bodily pain, health perceptions, physical, emotional, and social role functioning and mental health. Each item is scored on a 0 to 100 range, with a higher score indicating a worse outcome.
Short-Form NEURO-QoL | Change from baseline to 2-, 4-, 6-, 8-, 12-, 16-, and 20-weeks follow up visit
  Assesses quality of life related to neurological disorders. Each item ranges from 1-5, with a higher score indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Y Leung, MD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States